CLINICAL TRIAL: NCT02890680
Title: Randomized Double Blind Clinical Trial Evaluation of Bone Regeneration After Impacted Third Molar Surgery With the of Platelet-rich Fibrin: Pilot Study
Brief Title: Effects of the Use of Platelet-rich Fibrin on Bone Regeneration After Impacted Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, João Vitor dos Santos Canellas, DDS MS, MSc, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE 56621216.5.0000.5259
Record Dates: First submitted 2016-08-24; First posted 2016-09-07 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Fibrin/Therapeutic Use; Blood Platelets; Molar, Third; Bone Regeneration
Keywords: platelet-rich fibrin; third molar; bone regeneration
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platelet-rich fibrin group (Experimental): Use platelet-rich fibrin after mandibular third molar extraction
  Interventions: Procedure: Platelet-rich fibrin
- Control group (Placebo Comparator): mandibular third molar extraction
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Platelet-rich fibrin
  Arms: Platelet-rich fibrin group
Procedure: Control group
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the bone regeneration after impacted third molar surgery on split mouth design using platelet-rich fibrin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients
* Preoperative platelet count higher than 150,00/ mm3
* Patient who required bilateral mandibular third molar extractions

Exclusion Criteria:

* Smokers patients
* Alcoholics patients
* Patients whom the inferior second molar was missing
* Patients who had acute pericoronitis on the inferior third molar
* Severe periodontal disease

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in bone density through tomography evaluation | Change from Baseline bone measurement at three months after surgery

SECONDARY OUTCOMES:
Change in periodontal-probing depth measurement on distal aspect of the second molar through Clinical evaluation | Change from baseline at 3 months after surgery
Pain through Visual Analogue Scale | 1st day after surgery
Pain through Visual Analogue Scale | 3rd day after surgery
Pain through Visual Analogue Scale | 7th day after surgery
Soft tissue healing through Clinical evaluation numeric scale | 7th day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: João Vitor Canellas, DDS; MSc, Principal Investigator — Rio de Janeiro University State
Locations (1):
- João Canellas, Rio de Janeiro, Rio de Janeiro, Brazil